CLINICAL TRIAL: NCT00950482
Title: Pilot Study - The Impact of Traditional Acupuncture on Menopausal Vasomotor Symptoms, Psychological Stress and the Hypothalamic Pituitary Adrenal (HPA) - Sympathetic Nervous System (SNS) Axis: A Randomized, Controlled Trial
Brief Title: Pilot Study - Impact of Traditional Acupuncture on Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB# 16997
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Menopause
Keywords: Menopause; Acupuncture; Hotflash

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- TA (Active Comparator): Active TA
  Interventions: Procedure: TA
- AA (Active Comparator): Alternative Acupuncture
  Interventions: Other: AA
- WC (Active Comparator): Waiting Group
  Interventions: Other: WC

INTERVENTIONS:
Procedure: TA — In Traditional acupuncture (TA), in which eight acupuncture points are selected, subjects will undergo three 30-minute sessions weekly for 12 weeks. Disposable acupuncture needles (1-1.5 inch sterilized stainless steel)will be inserted up to one inch deep through a plastic needle tube that is secured with adhesive tape to the skin.
  Other Names: Traditional Acupuncture
  Arms: TA
Other: AA — In Alternative acupuncture (AA), in which eight acupuncture points are selected, subjects will undergo three 30-minute sessions weekly for 12 weeks. Disposable acupuncture needles (1-1.5 inch sterilized stainless steel)will be inserted up to one inch deep through a plastic needle tube that is secured with adhesive tape to the skin.
  Other Names: Alternative Acupuncture
  Arms: AA
Other: WC — Waiting Group
  Other Names: Waiting Group
  Arms: WC

SUMMARY:
This pilot project is a randomized research study to examine the effects of acupuncture on menopausal symptoms. The investigators will recruit up to 45 Cedars employees (excluding Dr Bairey Merz's employees) with menopausal symptoms by posting a study flyer on Exchange. If a patient is interested in this study, she may contact the research team for further information. Once a patient is identified as being eligible for the study, she will be contacted to schedule the screening visit. They will receive an explanation of the study. They will be sent the consent form to review prior to the initial visit. At the initial visit, prior to any study-related procedures, the consent will be reviewed with the patient. After all questions have been answered and the patient appears to fully understand the study, the patient will be asked to provide written consent.

This pilot project will collect data from three study groups as stated in the NIH application proposal. The first research study group will undergo traditional acupuncture (TA). The second research study group will receive alternative acupuncture (AA). The third group will be a waiting control group (WC) that will receive four weeks of acupuncture following completion of the study duration.

Traditional acupuncture means that the needle is inserted in true acupuncture point locations. Alternative acupuncture is a technique that varies slightly from traditional acupuncture and is used to assess which technique, if any, produces the best therapeutic results. Waiting control is a group of subjects who get neither traditional nor alternative acupuncture during the duration of treatment, which in this case, is 3 months.

Patients will be randomized into one of the three study groups, and will have one in three chance of being placed in one of the three groups. Neither patients nor the investigators can choose which group patients are assigned to. Patients from TA and AA groups will be asked to come to Cedars-Sinai a total of 39 times (36 sessions and 3 clinic visits) over a three-four month period. It will compare the effects (good or bad) of traditional acupuncture (TA) with alternative acupuncture (AA) on the menopausal symptoms to be studied in this research. Patients from WC group will be asked to come to Cedars-Siani a total of 15 times. Other study procedures include physical exam, blood and urine collection for hormone tests, questionnaire interview, etc.

During the pilot phase of this study subjects will record the number of mild, moderate, severe and/or very severe hot flashes that occur each day in a hot flash diary. There is also an option for patients to record other symptoms they may experience during that week other then hot flashes as well as a place for additional comments. Subjects will complete the diary for seven consecutive days. It is a simple form that takes very little time to complete each day (only 5-10 minutes) and will not impact the duration of the study participation.

No genetic study will be conducted in this pilot project.

DETAILED DESCRIPTION:
This pilot project is a randomized research study to examine the effects of acupuncture on menopausal symptoms. The investigators will recruit up to 45 Cedars employees (excluding Dr Bairey Merz's employees) with menopausal symptoms by posting a study flyer on Exchange. If a patient is interested in this study, she may contact the research team for further information. Once a patient is identified as being eligible for the study, she will be contacted to schedule the screening visit. They will receive an explanation of the study. They will be sent the consent form to review prior to the initial visit. At the initial visit, prior to any study-related procedures, the consent will be reviewed with the patient. After all questions have been answered and the patient appears to fully understand the study, the patient will be asked to provide written consent.

This pilot project will collect data from three study groups as stated in the NIH application proposal. The first research study group will undergo traditional acupuncture (TA). The second research study group will receive alternative acupuncture (AA). The third group will be a waiting control group (WC) that will receive four weeks of acupuncture following completion of the study duration.

Traditional acupuncture means that the needle is inserted in true acupuncture point locations. Alternative acupuncture is a technique that varies slightly from traditional acupuncture and is used to assess which technique, if any, produces the best therapeutic results. Waiting control is a group of subjects who get neither traditional nor alternative acupuncture during the duration of treatment, which in this case, is 3 months.

Patients will be randomized into one of the three study groups, and will have one in three chance of being placed in one of the three groups. Neither patients nor the investigators can choose which group patients are assigned to. Patients from TA and AA groups will be asked to come to Cedars-Sinai a total of 39 times (36 sessions and 3 clinic visits) over a three-four month period. It will compare the effects (good or bad) of traditional acupuncture (TA) with alternative acupuncture (AA) on the menopausal symptoms to be studied in this research. Patients from WC group will be asked to come to Cedars-Siani a total of 15 times. Other study procedures include physical exam, blood and urine collection for hormone tests, questionnaire interview, etc.

During the pilot phase of this study subjects will record the number of mild, moderate, severe and/or very severe hot flashes that occur each day in a hot flash diary. There is also an option for patients to record other symptoms they may experience during that week other then hot flashes as well as a place for additional comments. Subjects will complete the diary for seven consecutive days. It is a simple form that takes very little time to complete each day (only 5-10 minutes) and will not impact the duration of the study participation.

No genetic study will be conducted in this pilot project.

ELIGIBILITY:
Inclusion Criteria:

1. Women with menopausal Vasomotor symptoms (VMS) bothersome enough to warrant treatment;
2. Minimum of 7 hot flashes per day (on average);
3. Age limits: women ages 40-70 who have had at least one missed menstrual cycle or have undergone spontaneous menopause, women of any age who have medically induced menopause, women of any age who have had oophorectomy;
4. Informed written consent;
5. Ability to follow treatment protocols

Exclusion Criteria:

Exclusion Criteria (cohort):

1. Concomitant illness with reasonable likelihood of limiting survival to less than one year;
2. Current substance abuse (alcohol or drug);
3. Pregnancy known, suspected or planned in next year;
4. Non-English speaking patients
5. Men

Exclusion Criteria (TA intervention):

1. Other concomitant menopause treatment;
2. Participating in acupuncture treatment or formal psychological stress management program within the last year;
3. Participating in another treatment for VMS, unless willing to stop it 4 weeks in advance of participation;
4. HIV infection, chronic or active hepatitis or other blood-borne illness.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
vasomotor symptoms (VMS) frequency and severity | 3 months
  vasomotor symptoms (VMS) frequency and severity

SECONDARY OUTCOMES:
The Pittsburgh Sleep Diary (PghSD) | 60 minutes
Pittsburgh Sleep Quality Index (PSQI) | 30minutes
Beck Depression Inventory (BDI) | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Women's Heart Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Painovich JM, Shufelt CL, Azziz R, Yang Y, Goodarzi MO, Braunstein GD, Karlan BY, Stewart PM, Merz CN. A pilot randomized, single-blind, placebo-controlled trial of traditional acupuncture for vasomotor symptoms and mechanistic pathways of menopause. Menopause. 2012 Jan;19(1):54-61. doi: 10.1097/gme.0b013e31821f9171. PMID 21968279